CLINICAL TRIAL: NCT06592417
Title: To Evaluate the Phase I Clinical Study of JSKN016 in Chinese Patients With Advanced Malignant Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Alphamab Biopharmaceuticals Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JSKN016-101
Record Dates: First submitted 2024-04-28; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-04

CONDITIONS: Advanced Malignant Solid Tumor

STUDY DESIGN:
Intervention Model Description: Sequential Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dose escalation/expansion (Experimental): The subjects at dose escalation stage will be administered with investigational product (JSKN016) starting at 0.5 mg/kg, followed by1 mg/kg，2 mg/kg，4 mg/kg，6 mg/kg，7 mg/kg，8 mg/kgmg/kg, IV ,Q3W The subjects at dose expansion stage will be adiministered with JSKN016 at 6mg/kg or more(anticipated response dose)
  Interventions: Drug: JSKN016 injection

INTERVENTIONS:
Drug: JSKN016 injection — JSKN016 is a bispecific antibody drug conjugate targeting HER3 and TROP2.

SUMMARY:
This is a Phase I open, multi-center, first-in-human study evaluating JSKN016 in subjects with advanced metastatic solid tumors, divided into dose escalation and dose extension.

DETAILED DESCRIPTION:
A total of seven (Q3W, the first day of intravenous administration every 3 weeks) dose groups were designed during the dose escalation period. The dose groups were 0.5, 1.0, 2.0, 4.0, 6.0, 7.0 and 8.0 mg/kg, respectively. The DLT observation period was 21 days with accelerated titration BOIN design.

The specific steps for conducting a clinical trial using the BOIN design are as follows:

1. The accelerated titration is performed as follows: the first patient is assigned to dose level 1. If this patient does not develop dose-limiting toxicity (DLT), the second patient will be treated at the next higher dose level. Only one patient at a time is treated, and the dose-climbing process continues until the first DLT is observed, or a second grade 2 toxicity is present, or the highest dose is reached, or a Safety Inspection Committee (SMC) discussion decides to end accelerated titration, whichever occurs first. At least two more patients are then treated on the current dose. After that, follow steps 2 and 3 below with at least 3 patients in each group to treat follow-up patients (≥3 patients in the non-accelerated titration dose group).
2. Assign the dose to the next group of subjects according to the dose rise and fall rule shown in the Bayesian optimal interval (BOIN). Note the following:

   1. "Elimination" means the removal of current and higher doses from the trial. The removed dose is a hypertoxic dose and will no longer be used to treat any newly enrolled patients.
   2. If the current dose is removed, the dose is automatically lowered to the next lower level and administered to the subject for treatment. If the lowest dose is eliminated, the trial is terminated early to ensure subject safety. In this case, the MTD cannot be determined.
   3. If none of the decision conditions (i.e., raise, lower, or remove the dose) are met, continue to treat the next group (3 subjects) with the current dose.
   4. If the current dose is the minimum dose but the dose is still required to be reduced by the rules, the new subject is still treated at the current minimum dose. If the number of subjects with DLT reaches the exclusion threshold, the trial is terminated early to ensure subject safety.
   5. If the current dose is the maximum dose but a higher dose is required by rule, the new subject is treated at the current maximum dose.
3. Repeat Step 2 until the set dose escalation phase has a maximum sample size of 20, or the number of evaluable subjects treated at the current dose reaches 9 and the current decision is to maintain the current dose according to the rise and fall rule of the dose escalation decision table.

During dose escalation, the SMC will conduct an ongoing safety assessment. The safety data for each dose group is reviewed by the SMC before the next dose group is administered. For the 6th dose group 7 mg/kg, SMC can decide whether to skip this dose group by comprehensively considering the previous safety, PK and other data. The composition and responsibilities of the SMC will be further detailed in the SMC Constitution.

In each dose group, the administration of the second subject was initiated at least 24 hours after the administration of the first subject to identify some acute toxicities, such as infusion-related reactions.

Allow patients to proceed with intragroup dose escalation to minimize the potential for undertreatment of patients. Intrapatient dose escalation will be performed in the following manner: (1) Intrapatient dose escalation will only be performed if ≤ grade 2 toxicity is observed during the previous treatment cycle; (2) Does not increase to the next higher dose level until the full DLT observation period is evaluated for the next higher dose level and the SMC does not confirm safety concerns; (3) Patients receiving the first dose escalation should be dosed for at least 4 cycles without disease progression. For example, if patients in the 1 mg/kg group completed DLT observation and 4 cycles of dosing, only if patients in the 2 mg/kg cohort completed a complete DLT evaluation, the SMC did not confirm safety concerns, and no grade 2 toxicity was observed in patients in the 1 mg/kg cohort during the previous treatment cycle. Subsequent doses may be increased to 2 mg/kg with the consent of the SMC.

The recommended dose for cohort expansion (RDE) will be determined by the SMC based on safety/tolerability, PK data, and preliminary antitumor activity, as well as other available data. RDE can be at the same dose level as MTD or at a lower dose level than MTD; Rdes may also be different for different indications.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subjects can understand the informed consent form, voluntarily participate in and sign the informed consent form; 2. The subjects were ≥18 years old on the day of signing the informed consent, male or female; 3. Subjects with histologically and/or cytologically confirmed advanced unresectable or metastatic epithelial malignancies that have failed or are intolerable to previous standard therapies, preferentially but not limited to the following types: AGA-positive non-small cell lung cancer, HER2 IHC 0 breast cancer, etc.

  4. For AGA-positive NSCLC, the presence of at least one of the following mutations is required; EGFR, ALK, ROS1, NTRK, BRAF V600, MET exon 14, RET, KRAS G12C, or HER2;
  * For the enrolled subjects, the above driver gene mutations were not tested, but the previous test results confirmed by the investigators were accepted;
  * If only EGFR overexpression without driver gene mutation can not be included;
  * Prior osimertinib therapy is required if EGFR T790M mutation is present;
  * Participants had to have failed at least one prior targeted therapy and at least platinum-based chemotherapy with or without an immune checkpoint inhibitor or antiangiogenic agent; 5. Breast cancer patients with HER2 IHC 0 expression, regardless of hormone receptor (HR) expression, could be enrolled according to the results of IHC examination in our center.

    6. At least one measurable lesion at baseline according to RECIST 1.1 criteria. Measurable disease required either no previous local treatment (e.g., radiotherapy) or evidence of disease progression after local treatment.

    7. Expected survival time ≥3 months; 8. ECOG score 0 or 1; 9. Female subjects of childbearing potential or male subjects with a fertile partner agreed to use highly effective contraception from the time they provided written informed consent until 24 weeks after the last dose. Female subjects of childbearing potential had to have a negative serum/urine pregnancy test within 7 days before randomization (for women of childbearing age, see Appendix 2).

    10. Adequate organ function within 7 days before randomization:
  * Bone marrow function: absolute neutrophil count ≥1.5×109/L; Hemoglobin ≥90 g/L; Platelet count ≥100×109/L (no whole blood or blood component transfusion within 14 days before randomization; No administration of hematopoietic cytokines within 7 days before randomization).
  * Liver function (based on the normal value of each clinical research center) : total bilirubin < 1.5 times the upper limit of normal value (ULN, total bilirubin in subjects with liver metastasis ≤3 x ULN); ALT/AST≤3×ULN (≤5×ULN in patients with liver metastasis); Albumin ≥28g/L; Renal function: serum creatinine ≤1.5 times the upper limit of normal, or creatinine clearance (Ccr) calculated according to Cockcroft-Gault formula (see Appendix 4) ≥ 60 mL/min; Coagulation function: INR or PT≤ 1.5x ULN, and aPTT≤ 1.5x ULN (low stable dose of anticoagulant, such as aspirin 100 mg/ day is allowed); 11. Left ventricular ejection fraction (LVEF) ≥50% (by echocardiography [ECHO]); 12. Participants were able and willing to comply with protocol-specified visits, treatment plans, laboratory tests, and other study-related procedures.

Exclusion Criteria:

* 1. Patients with symptoms of active central nervous system metastases, except those with stable parenchymal brain metastases as assessed by investigators, were defined as seizure-free for more than 12 weeks with or without the use of antiepileptic drugs; No need for glucocorticoids; At least one MRI showed that the patient was stable on imaging. Or stable after treatment for more than 1 month without symptoms; 2. Received any investigational drug within 28 days before dosing; 3. Receipt of other antineoplastic therapy within 28 days before dose or within 5 half-lives of previous antineoplastic drugs, whichever is shorter but requires a minimum of 14 days; Received Chinese herbal medicine with clear anti-tumor indications within 14 days before drug administration; 4. Local palliative treatment within 14 days before administration; 5. Major surgical treatment (such as transabdominal or transthoracic surgery) within 28 days before drug administration; Excluding minor procedures such as diagnostic punctures or infusion device implantation or biliary stenting) or anticipated need for major surgical treatment during the study period; 6. Gastrointestinal abnormalities with obvious clinical manifestations, including but not limited to: intestinal obstruction or the presence of symptoms and signs of intestinal obstruction within 6 months before drug administration, but if the obstruction was completely removed after surgical treatment, screening could be performed (patients with previous intestinal stent implantation and the intestinal stent was not removed during the screening period were not allowed); Patients with gastrointestinal perforation, gastrointestinal fistula, intra-abdominal abscess and non-gastrointestinal fistula (such as tracheoesophageal fistula) within 6 months before administration; Patients with gastrointestinal bleeding (CTCAE≥ grade 3) within 6 months before treatment, or gastrointestinal bleeding (melena, bloody stool, etc.) within 1 month before randomization were eligible if hemorrhoid bleeding was confirmed or only showed positive fecal occult blood.

  7. Subjects with uncontrolled massive serous effusion or moderate to massive serous effusion requiring repeated drainage (recurrence within 2 weeks after intervention) such as pleural effusion, pericardial effusion, ascites, cachexia, etc.

  8. Always received including the antibody coupling of topoisomerase inhibitors class I drug therapy, such as DS-8201, HER3-DXd, DS-1062, etc; 9. A history of (noninfectious) interstitial lung disease (ILD) or noninfectious pneumonia requiring steroid therapy, current ILD or noninfectious pneumonia, or ILD or noninfectious pneumonia that could not be ruled out by imaging at screening; 10. Other malignant tumors within 5 years before drug administration, Cured cutaneous squamous cell carcinoma, basal cell carcinoma, non-primary invasive bladder cancer (defined as stage ≤T2a, Gleason score ≤6, and at the time of prostate cancer diagnosis) were excluded Patients with PSA≤10ng/mL (if measured) who had received radical treatment and had no PSA biochemical recurrence could participate in the study), in situ prostate/cervix/breast cancer; 11. Have uncontrolled comorbidities, including but not limited to the following:
* Active HBV or HCV infection Patients with HBsAg (+) and HBV-DNA< 2500 copies /mL or 500 IU/mL were allowed to be enrolled. HCV-Ab (+) and HCV-RNA negative were allowed to enroll.

  * HIV infection;
  * Known active tuberculosis; Active syphilis;
  * Active or uncontrolled infection requiring systemic anti-infective treatment; Uncontrolled hypertension (systolic blood pressure ≥160mmHg, Diastolic blood pressure > 100 mmHg), symptomatic heart failure (NYHA II-IV), unstable angina or myocardial infarction within 6 months, history of heart failure or systolic dysfunction (LVEF<50%), or risk of QTc prolongation or arrhythmia (baseline QTc>470 msec) ), intractable hypokalemia, long QT syndrome, tachycardia at rest with a heart rate >100 bpm, atrial fibrillation or clinically symptomatic valvular heart disease (if well controlled by treatment), moderate-severe pulmonary hypertension, or a history of other arrhythmias of medical importance).

Newly diagnosed thromboembolic events requiring treatment within 6 months (patients with well-controlled deep-vein thrombosis of the lower extremities or venous access ports were allowed).

12. The toxicity of previous antineoplastic therapy did not recover to CTCAE grade ≤1 (NCI-CTCAE v5.0); Note: Subjects with stable CTCAE grade 2 toxicity related to previous antineoplastic therapy (defined as stable toxicity severity and no CTCAE grade greater than 2 within 3 months before dose administration) could be enrolled, such as: Chemotherapy-induced neurotoxicity, alopecia, skin pigmentation, fatigue, endocrine toxicity caused by previous immunotherapy (such as thyroid dysfunction, diabetes, hyperglycemia, adrenal insufficiency); 13. Previous history of allogeneic bone marrow or organ transplantation; 14. Previous history of allergic reaction or anaphylaxis to antibody drugs; 15. Previous history of severe dry eye, severe meibomian gland disease and/or blepharitis, keratopathy and maculopathy resulting in untreatable or delayed corneal healing of the subject; 16. Pregnant and/or lactating women; 17. Other conditions considered by the investigators to affect the safety or compliance of the study drug treatment, including but not limited to mental disorders, alcohol or drug abuse, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-05-17 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of DLTs | 21 days after the first dose for subjects at dose escalation stage
  DLTs are defined as one or more serious toxic reactions that occur within 21 days (Q3W) after the start of dosing and are determined to be reasonably associated with the study drug
The frequency and severity of treatment-related adverse events (TEAE), treatment-related adverse events (TRAE), and serious adverse events (SAE). | From first dose to 30 days after last dose
  Clinically significant changes in lab test findings
MTD or RP2D of JSKN 016 | Postdose of last participant up to 1 year
  To determinate MTD and/ or RP2D of JSKN016
Objective Response Rate (ORR) in Extended queue | Postdose of last participant up to 1 year
  Objective response rate (ORR) was defined as the proportion of participants who achieve either complete response [CR] or partial response [PR] per Response Evaluation Criteria in Solid Tumors (RECIST v1.1）

SECONDARY OUTCOMES:
Clinical benefit rates (CBR) | Postdose of last participant up to 1 year
  Clinical benefit rate (CR+PR+[stable disease (SD) ≥ 6 months]) is defined as those participants with best response as CR or PR or else SD with a duration of at least 6 months. SD for 6 months duration was defined as the time from the first dose to the first documentation of PD or to the last adequate response assessment prior to data cut-off date, whichever is earlier.
Cmax of JSKN016 | Predose to 90 days after last dose
  Maximum (Peak) Observed blood Concentration (Cmax) of JSKN016 Following First Dose
Tmax of JSKN016 | Predose to 90 days after last dose
  Time of Maximum blood Concentration (Tmax) of JSKN016 Following First Dose
AUC of JSKN016 | Postdose of last participant up to 1 year
  The blood PK parameters of JSKN016 and its analytes for area under the concentration-versus-time curve from time 0 to the last quantifiable concentration as calculated by the linear-up log-down trapezoidal method (AUClast) and AUC from time 0 to infinity (AUCinf) elimination rate constant associated with the terminal phase were estimated using standard non-compartmental methods.
Terminal Elimination Half-life (t1/2) | Postdose of last participant up to 1 year
  The blood PK parameters of Terminal elimination half-life for JSKN016
Duration Of Response (DOR) | Postdose of last participant up to 1 year
  Defined as the time from the first evaluation of objective response to the first evaluation of PD or death from any cause prior to PD

CONTACTS AND LOCATIONS:
Overall Officials: Jieqiong Liu, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (2):
- China (2):
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Hospital, Sun Yat-sen University, Guangzhou, Guangdong

IPD SHARING:
Plan to Share IPD: No